CLINICAL TRIAL: NCT04942340
Title: Turning Dexmedetomidine Into a Powerful Anesthetic That Can be Rapidly and Completely Reversed
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Withdrawn secondary to a change in protocol design forthcoming.
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB21-0922
Record Dates: First submitted 2021-06-11; First posted 2021-06-28 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Emergence From Anesthesia
Keywords: Atipamezole; Caffeine; Sedation Recovery; Anesthesia; Precedex
MeSH Terms: interventions — atipamezole; Caffeine; Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: TBA
Who Masked: Investigator
Masking Description: The anesthesiologists will be blinded to the medication injected to the subject since the drugs or normal saline are prepared by the pharmacists in the OR pharmacy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase 1: Atipamezole & caffeine's in a 1:1 ratio (Active Comparator): Is this arm, subjects will be randomized to IV administration of Atipamezole & caffeine's in a 1:1 ratio
  Interventions: Drug: Atipamezole & Caffeine
- Phase 1: Precedex & Saline in a 1:1 ratio (Placebo Comparator): Is this arm, subjects will be randomized to receive IV administration of Precedex & Saline in a 1:1 ratio
  Interventions: Drug: Dexmedetomidine Hydrochloride & Saline

INTERVENTIONS:
Drug: Atipamezole & Caffeine — In this arm, subjects will be infused with Atipamezole (2 g/kg) and caffeine (15 mg/kg) across 5 minutes
  Other Names: Antisedan
  Arms: Phase 1: Atipamezole & caffeine's in a 1:1 ratio
Drug: Dexmedetomidine Hydrochloride & Saline — In this arm, subjects will be infused with Precedex & Saline at 15 mg/kg across 5 minutes
  Other Names: Precedex
  Arms: Phase 1: Precedex & Saline in a 1:1 ratio

SUMMARY:
In this study, the investigators will explore Atipamezole & caffeine's ability to facilitate the emergence from anesthesia. Each subject will visit UChicago 4 times. The first time for informed consent. The second time for a complete physical exam to ensure that the subjects are healthy. Then there are 2 sedation sessions. Subjects get an honorarium for each sedation session.

DETAILED DESCRIPTION:
Each subject will attend 3 sessions to complete the study. In the first session, an anesthesiologist will take a medical history and perform a physical examination on the subject. A baseline EKG and urine drug screen test will be obtained. If the subject meets the criteria for the study, healthy and drug-free, the risks involved in the study will be covered in detail. If the subject is willing, then that subject will be enrolled in the study and a detailed informed consent form will covered in detail. Prior to signing the consent form the subject will be required to describe the risks involved in the study in their own words, showing that each subject understand. For each session, subjects will be asked not to eat and drink 8 hours prior to the study in order to minimize the potential risk for aspiration during anesthesia

Once the subject is checked in, a peripheral intravenous catheter (IV) will be inserted on one of the arms. A second IV will be inserted to the other arm. After the IV insertion, American Society of Anesthesiologists (ASA) standard monitoring, including EKG, blood pressure (BP), respiratory rate, pulse oximetry and temperature, will be used to assess the subject. An EEG monitor probe will be applied to the forehead skin as well. The subject will then be asked to breathe 100% reof Precedex (2 g/kg), via pump, across 10 minutes. There will be a 5 minute interval to allow the drug to equilibrate. Then p or saline (control). The face mask will stay in place throughout the procedure. For the experiment described, Ati: Dex ratio is 1:1. The investigators will be blind to the injection.

The investigators will measure the time when the drug injections are complete to the awakening of the subject. The investigators will record the time until the subject's eyes open, and the time until the subject can respond to the command to grip the hand of the attending physician. When the subject is awake and alert (oriented to time, place and name), the subject will perform psychomotor tests to measure his cognitive function. The subject will be required to complete a simple set of cognitive tests to determine if they are still impaired by the sedative. Both "control" and test subjects will be required to complete the same tests. Tests include one for hand-eye coordination by tracking a randomly moving circle on a computer screen with a cross controlled by a mouse. Reaction time is measured by asking the subject to press a button when the subject hears a sound. The tests will be repeated every 15 minutes for 90 minutes after waking. This will allow the investigators to get a recovery time course.

ELIGIBILITY:
Inclusion Criteria:

1. Age >21 or <40
2. ASA physical status = 1 (normal healthy patient without systematic diseases or conditions)
3. Metabolic Equivalents of Functional Capacity (METs) > 5
4. Low risk for Obstructive Sleep Apnea (OSA) based on the screening test (STOP-bang score established by American Society of Sleep Apnea): Yes to < 3 items- high risk of OSA
5. No history Arrhythmia, such as heart block (Baseline EKG will be obtained during the history and physical session), seizure, liver and kidney diseases
6. BMI <30 kg/m2
7. No history of any mental illness
8. No history of drugs or alcohol abuse (an urine drug screen test required)

Exclusion Criteria:

1. Age <21 or >40
2. ASA physical status > 1 (normal healthy patient with systematic diseases or conditions)
3. Metabolic Equivalents of Functional Capacity (METs)<5
4. High risks for Obstructive Sleep Apnea (OSA) based on the screening test (STOP-bang score established by American Society of Sleep Apnea): Yes to > 3 items- high risk of OSA
5. History Arrhythmia (Baseline EKG will be obtained during the history and physical session), seizure, liver and kidney diseases
6. BMI >30 kg/m2
7. History of any mental illness
8. History of drugs or alcohol abuse (an urine drug screen test required)
9. Female subjects with positive urine pregnancy test, which will be performed before each sedation session

Ages: 22 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
The time when the drug injections are complete to the awakening of the subject. | 1 Day
  We will record the time until the subject's eyes open, and the time until the subject can respond to the command to grip the hand of the attending physician

SECONDARY OUTCOMES:
Measure Cognitive Function | This test will be repeated every 15 Minutes for 90 Minutes after the subject has awakened]
  Subjects will be asked to track randomly moving circle on a computer screen with a cross controlled by a mouse
Measure Reaction Time | This test will be repeated every 15 Minutes for 90 Minutes after the subject has awakened]
  Subjects will be asked to press a button when he/ she hears a sound

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided